CLINICAL TRIAL: NCT04619992
Title: Consumer Evaluation of Intermittent Catheter Product Modifications
Status: Completed | Type: Interventional
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6009-CONT
Record Dates: First submitted 2020-10-27; First posted 2020-11-06 (Actual); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Urinary Incontinence
Keywords: Intermittent Catheterization
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Current users of Hollister standard with tip hydrophilic intermittent catheters (Other): Subjects in this arm are current users of Hollister standard with tip hydrophilic intermittent catheters.
  Interventions: Device: Test Hydrophilic Intermittent Catheter
- New users of Hollister standard with tip hydrophilic intermittent catheters (Other): Subjects in this arm are new users of Hollister standard with tip hydrophilic intermittent catheters.
  Interventions: Device: Currently marketed Hydrophillic Intermittent Catheter; Device: Test Hydrophilic Intermittent Catheter

INTERVENTIONS:
Device: Currently marketed Hydrophillic Intermittent Catheter — Currently marketed Hollister standard with tip hydrophilic intermittent catheter
  Arms: New users of Hollister standard with tip hydrophilic intermittent catheters
Device: Test Hydrophilic Intermittent Catheter — Hollister standard with tip hydrophilic intermittent catheter with design enhancements

SUMMARY:
This study aims to collect feedback from hydrophilic intermittent catheter end-users to assess user acceptance of the test hydrophilic intermittent catheter and generate evidence to support commercial marketing objectives.

ELIGIBILITY:
A. Inclusion Criteria for Arm 1

Subject who:

1. is male and at least 18 years of age
2. has been performing unassisted, self-catheterizations, with a Hollister standard with tip Hydrophilic intermittent catheter, 3 or more times a day for at least 1 month

B. Exclusion Criteria for Arm 1

Subject who:

1. is currently undergoing chemotherapy, radiation or steroid therapy
2. has a symptomatic urinary tract infection (UTI)
3. is currently using a coude intermittent catheter product to perform catheterization
4. performs non-urethral catheterization

C. Inclusion Criteria for Arm 2

Subject who:

1. is male and at least 18 years of age
2. has been performing unassisted, self-catheterizations, with a non-standard with tip Hydrophilic intermittent catheter, 3 or more times a day for at least 1 month

D. Exclusion Criteria for Arm 2

Subject who:

1. is currently undergoing chemotherapy, radiation or steroid therapy
2. has a symptomatic urinary tract infection (UTI)
3. is currently using a coude intermittent catheter product to perform catheterization
4. performs non-urethral catheterization
5. is unable to use a Hollister standard with tip hydrophilic intermittent catheter

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hollister Incorporated, Libertyville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Current Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters | New Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters
Started | 55 | 7
Completed | 54 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Current Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters | New Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters | Total
Number analyzed (Participants) | 54 | 7 | 61
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  18-29 years | 8 | 0 | 8
  30-39 years | 12 | 0 | 12
  40-49 years | 11 | 1 | 12
  50-59 years | 10 | 2 | 12
  60-69 years | 9 | 1 | 10
  70-79 years | 3 | 3 | 6
  80-89 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Per protocol inclusion criteria, only males were eligible for participation.
  Participants
    Female | 0 | 0 | 0
    Male | 54 | 7 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 54 | 7 | 61

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Test Hydrophilic Intermittent Catheter
Description: Users will rate if Test device is an acceptable alternative to currently marketed device. Acceptability will be rated via a standard 5-point Likert agreement scale. Agreement signifies Test catheter is an acceptable alternative to currently marketed catheter.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Current Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters | New Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters
Number analyzed (Participants) | 54 | 7
Participants
  'Strongly agree' or 'Agree' | 45 | 4
  Neither agree nor disagree | 4 | 2
  'Disagree' or 'Strongly disagree' | 5 | 1

2. Primary Outcome: Preference of Test Hydrophilic Intermittent Catheter
Description: Users will rate if Test device is preferred to currently marketed device. Preference will be rated via a standard 5-point Likert agreement scale. Agreement signifies Test catheter is preferred to currently marketed catheter.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Current Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters | New Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters
Number analyzed (Participants) | 54 | 7
Participants
  'Strongly agree' or 'Agree' | 35 | 4
  Neither agree nor disagree | 11 | 2
  'Disagree' or 'Strongly disagree' | 8 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the duration of the study (October 2020 to August 2021), an average of 12 days per subject.
Arm/Group | Current Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters | New Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/7
Other Adverse Events (participants affected / at risk) | 7/54 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Current Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters (N=54) | New Users of Hollister Standard With Tip Hydrophilic Intermittent Catheters (N=7)
Potential viral infection (Infections and infestations) | 1 (1) | 0 (0) — Probably not related to study product. Mild severity. Subject reported increased fatigue and muscular aches. Undiagnosed but most likely due to viral infection. No urinary tract infection present. Self-resolved after few days.
Ankle surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Unrelated to study product. Mild severity. Subject underwent ankle surgery.
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated to study product. Mild severity. Subject reported loose stools. Self-resolved after few days.
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Probably not related to study product. Moderate severity. Subject undergoing bowel management program. History of urinary tract infections during bowel training.
Urethral discomfort (Product Issues) | 0 (0) | 1 (1) — Possibly related to study product. Mild severity. Burning sensation while inserting urinary catheter for initial insertions. No other urinary or product complications present.
Cloudy urine (Renal and urinary disorders) | 1 (1) | 0 (0) — Probably not related to study product. Mild in severity. Subject reports cloudy urine. Resolved after 48 hours. No other urinary complications present.
Reduced urine flow and hip spasticity (Renal and urinary disorders) | 1 (1) | 0 (0) — Possibly related to study product. Mild in severity. Subject reported sensation of incomplete bladder voiding and hip spasticity. Improper storage of study product led to potential kinking of catheter tube. Issue resolved after proper storage.
Potential urethral narrowing (Renal and urinary disorders) | 1 (1) | 0 (0) — Unrelated to study product. Moderate severity. Subject had difficulty inserting catheter due to potential urethral narrowing. This complication was present prior to use of study product and under the care of healthcare provider.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT04619992/Prot_SAP_001.pdf